CLINICAL TRIAL: NCT03814447
Title: The Clinical Research of Fourth Generation CART-cell Therapy in Refractory-Relapsed Ovarian Cancer
Brief Title: The Fourth Generation CART-cell Therapy for Refractory-Relapsed Ovarian Cancer
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai 6th People's Hospital (Other)
Collaborators: Hrain Biotechnology Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Zhao Hui, professor, Shanghai 6th People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MESO-CART
Record Dates: First submitted 2019-01-18; First posted 2019-01-24 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Ovarian Cancer
Keywords: MESO; CAR-T; Ovarian cancer; Refractory-Relapsed
MeSH Terms: conditions — Ovarian Neoplasms | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti- MESO CAR-T cells (Experimental): The subjects in this arm will receive Cyclophosphamide 300mg/m2/d and Fludarabine 30mg/m2/d d-4~-2. Then anti- MESO CAR-T cells will be injected by a dose of 5×106/kg once at d1(rang from d1-3).
  Interventions: Drug: anti- MESO CAR-T cells; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: anti- MESO CAR-T cells — Autologous genetically modified anti- MESO CAR transduced T cells
Drug: Fludarabine — Dose: 30mg/m2/d
  Other Names: FA
Drug: Cyclophosphamide — Dose: 300mg/m2/d
  Other Names: CTX

SUMMARY:
The goal of this clinical trial is to study the safety and feasibility of anti- Mesothelin Chimeric Antigen Receptor T-Cell (MESO CAR-T cells) therapy for Refractory-Relapsed Ovarian Cancer

DETAILED DESCRIPTION:
Primary Objectives:

1. To determine the safety and feasibility of anti- MESO CAR-T cells therapy for Refractory-Relapsed Ovarian Cancer

Secondary Objectives:

1. To access the efficacy of anti- MESO CAR-T cells in patients with ovarian cancer.
2. To determine in vivo dynamics and persistency of anti- MESO CAR-T cells
3. To assess the quality of life in patients with ovarian cancer after treatment with anti- MESO CAR-T cells.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically confirmed ovarian cancer;
2. 18-75 Years Old, female;
3. Expected survival > 12 weeks;
4. Eastern Cooperative Oncology Group (ECOG) score 0-2;
5. Patients who have previously been treated with second- line or above standard treatment are failed (progress in treatment or recurrence within 6 months after discontinuation of treatment);
6. According to the Immune-Modified Response Evaluation Criteria In Solid Tumors (imRECIST) , there should be at least one measurable tumor foci；
7. Positive expression of Mesothelin in tumor tissue；
8. Creatinine ≤ 1.5×ULN or creatinine clearance ≥ 60ml / min;
9. alanine aminotransferase and aspartate aminotransferase ≤ 2.5×ULN , such as with liver metastasis, ≤ 5×ULN;
10. Total bilirubin ≤ 2×ULN;
11. Hemoglobin≥90g/L(No blood transfusion within 14 days);
12. Absolute value of neutrophils ≥1.5×10^9/L;
13. Absolute counting of lymphocytes >0.7×10^9/L;
14. Counting of Platelet≥80×10^9/L；
15. The venous access required for collection can be established without contraindications for leukocyte collection;
16. Able to understand and sign the Informed Consent Document.

Exclusion Criteria:

1. Accompanied by other uncontrolled malignant tumors;
2. Active hepatitis B, hepatitis C, syphilis, HIV infection;
3. Insufficient function of important organs (heart, lung);
4. Any other uncontrolled active disease that impedes participation in the trial;
5. Any affairs could affect the safety of the subjects or purpose this trial;
6. Pregnant or lactating women, or patients who plan to be pregnancy during or after treatment;
7. There are active or uncontrollable infections (except simple urinary tract infections or upper respiratory tract infections) that require systemic therapy within 14 days or 14 days prior to enrollment；
8. The investigator believes that it is not appropriate to participate in the trial;
9. Received CAR-T treatment or other gene therapies before enrollment; Subjects suffering disease affect the understanding of informed consent or unable to comply with study; Unwilling or unable to comply with study requirements.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-08-16 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) and Serious adverse event (SAEs) | 1 year post infusion
  Safety measured by occurrence of study related adverse effects defined by NCI CTCAE 4.03

SECONDARY OUTCOMES:
Cmax | 30 days post infusion
  the highest concentration (Cmax) of anti-human MESO T cells in the peripheral blood after administration
Tmax | 30 days post infusion
  the time to reach the highest concentration (Tmax) of anti-human MESO T cells in the peripheral blood after administration
AUC(0-30d) | 30 days post infusion
  the area under the curve of 30 days of anti-human MESO T cells in the peripheral blood after administration
Duration of Mesothelin-positive T cells in circulation | 90 days post infusion
  Duration of Mesothelin-positive T cells in circulation
ORR | 3 months post infusion
  Overall response rate after administration
PFS | 1 year post infusion
  Progress Free Survival after administration
EORTC Quality-of-Life Questionnaire Core 15 Palliative Care (QLQ-C15-PAL) of patients after administration | 1 year post infusion
  This QLQ-C15-PAL score consists of 15 questions; two multi-item functional scales (physical and emotional functioning), two multi-item symptom scales (fatigue and pain) together with five single-item symptom scales (nausea/vomiting, dyspnea, insomnia, appetite loss, constipation) and one final question referring to overall QOL. The physical functioning scale is based on three questions regarding walking, activities of daily living and time spent in bed or in a chair. The emotional functioning scale is based on two questions that ask about feeling tense or depressed. Patients rated each question on a Likert scale from 1 (not at all) to 4 (very much), with the exception of overall QOL, which was rated from 1 (very poor) to 7 (excellent)

CONTACTS AND LOCATIONS:
Overall Officials: Hui Zhao, doctor, Principal Investigator — Shanghai 6th People's Hospital
Locations (1):
- Shanghai 6th People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No